CLINICAL TRIAL: NCT06809387
Title: Investigating the Supplementary Motor Area Role in Speech and Reading Fluency in PWS With rTMS
Brief Title: Investigating the SMA's Role in Speech and Reading Fluency in PWS With rTMS
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Gülkader Temiz, Principal Investigator, Medipol University
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: E-10840098-202.3.02-645
Record Dates: First submitted 2024-11-26; First posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2024-11

CONDITIONS: Stuttering, Adult
Keywords: rTMS; stuttering; SMA
MeSH Terms: conditions — Stuttering | interventions — Deep Brain Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Real rTMS (Experimental): Participants will be included in the real rTMS. Participants will perform speech and reading tasks before and after stimulation.
  Interventions: Other: Brain stimulation
- Sham rTMS (Placebo Comparator): Participants will be included in the sham rTMS. Participants will perform speech and reading tasks before and after stimulation.
  Interventions: Other: Brain stimulation

INTERVENTIONS:
Other: Brain stimulation — Participants will be included in the real and sham rTMS. Participants will perform speech and reading tasks before and after stimulation.

SUMMARY:
The goal of this clinical trial is to study how a part of the brain called the supplementary motor area (SMA) is connected to speech and reading fluency in adults who stutter. Researchers will use a method called repetitive transcranial magnetic stimulation (rTMS) to learn more about this relationship. The main question it aims to answer is:

-Will participants' speech and reading fluency improve when we stimulate the SMA with rTMS?

Participants will take part in both placebo rTMS and real rTMS sessions.

Participants will:

* Come to the research center for 2 days, with at least a one-week break between visits
* Read 4 passages and speak on 4 topics
* Be video recorded while doing these tasks

ELIGIBILITY:
Inclusion Criteria:

* To be over 18 years of age
* Presence of developmental stuttering
* Being right hand dominant

Exclusion Criteria:

* Being under 18 years of age
* The presence of a diagnosed brain lesion
* Presence of intracranial metal implantation
* Presence of a speech and language problem other than stuttering
* The presence of a diagnosed neurological disorder
* The presence of a diagnosed psychiatric disorder
* Use of drugs and substances that may affect the central nervous system
* History of epilepsy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-06-15 (Estimated); Study Completion 2025-06-15 (Estimated)

PRIMARY OUTCOMES:
Severity of stuttering in speech and reading Day 1 (pre-treatment) | Immediately before the treatment (Day 1)
  Stuttering severity will be calculated on video recordings taken during speaking and reading tasks. Stuttering Severity Instrument - 4th Edition (SSI-4) scale will be used for this.
Severity of stuttering in speech and reading Day 1 (post-treatment) | Immediately after the treatment (Day 1)
  Stuttering severity will be calculated on video recordings taken during speaking and reading tasks. Stuttering Severity Instrument - 4th Edition (SSI-4) scale will be used for this.
Severity of stuttering in speech and reading Day 2 (pre-treatment) | Immediately before the treatment (Day 2)
  Stuttering severity will be calculated on video recordings taken during speaking and reading tasks. Stuttering Severity Instrument - 4th Edition (SSI-4) scale will be used for this.
Severity of stuttering in speech and reading Day 2 (post-treatment) | Immediately after the treatment (Day 2)
  Stuttering severity will be calculated on video recordings taken during speaking and reading tasks. Stuttering Severity Instrument - 4th Edition (SSI-4) scale will be used for this.

CONTACTS AND LOCATIONS:
Locations (1):
- İstanbul Medipol Üniversitesi Dil, Konuşma ve Yutma Terapisi ve Yenilikçi Teknolojiler Merkezi (MEDKOM), Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP
Time Frame: January 2025-January 2026

REFERENCES:
- [Background] Wassermann EM. Risk and safety of repetitive transcranial magnetic stimulation: report and suggested guidelines from the International Workshop on the Safety of Repetitive Transcranial Magnetic Stimulation, June 5-7, 1996. Electroencephalogr Clin Neurophysiol. 1998 Jan;108(1):1-16. doi: 10.1016/s0168-5597(97)00096-8. PMID 9474057
- [Background] Tezel-Bayraktaroglu O, Bayraktaroglu Z, Demirtas-Tatlidede A, Demiralp T, Oge AE. Neuronavigated rTMS inhibition of right pars triangularis anterior in stuttering: Differential effects on reading and speaking. Brain Lang. 2020 Nov;210:104862. doi: 10.1016/j.bandl.2020.104862. Epub 2020 Sep 23. PMID 32979643
- [Background] Rossi S, Hallett M, Rossini PM, Pascual-Leone A; Safety of TMS Consensus Group. Safety, ethical considerations, and application guidelines for the use of transcranial magnetic stimulation in clinical practice and research. Clin Neurophysiol. 2009 Dec;120(12):2008-2039. doi: 10.1016/j.clinph.2009.08.016. Epub 2009 Oct 14. PMID 19833552
- [Background] Neef NE, Anwander A, Friederici AD. The Neurobiological Grounding of Persistent Stuttering: from Structure to Function. Curr Neurol Neurosci Rep. 2015 Sep;15(9):63. doi: 10.1007/s11910-015-0579-4. PMID 26228377
- [Background] Etchell AC, Civier O, Ballard KJ, Sowman PF. A systematic literature review of neuroimaging research on developmental stuttering between 1995 and 2016. J Fluency Disord. 2018 Mar;55:6-45. doi: 10.1016/j.jfludis.2017.03.007. Epub 2017 Mar 12. PMID 28778745
- [Background] Busan P, Del Ben G, Russo LR, Bernardini S, Natarelli G, Arcara G, Manganotti P, Battaglini PP. Stuttering as a matter of delay in neural activation: A combined TMS/EEG study. Clin Neurophysiol. 2019 Jan;130(1):61-76. doi: 10.1016/j.clinph.2018.10.005. Epub 2018 Nov 10. PMID 30476712
- [Background] Busan P. Developmental stuttering and the role of the supplementary motor cortex. J Fluency Disord. 2020 Jun;64:105763. doi: 10.1016/j.jfludis.2020.105763. Epub 2020 Apr 20. PMID 32361030
- [Background] Brown S, Ingham RJ, Ingham JC, Laird AR, Fox PT. Stuttered and fluent speech production: an ALE meta-analysis of functional neuroimaging studies. Hum Brain Mapp. 2005 May;25(1):105-17. doi: 10.1002/hbm.20140. PMID 15846815
- [Background] Alm PA. Stuttering and the basal ganglia circuits: a critical review of possible relations. J Commun Disord. 2004 Jul-Aug;37(4):325-69. doi: 10.1016/j.jcomdis.2004.03.001. PMID 15159193